CLINICAL TRIAL: NCT02677298
Title: Randomized Double Blind Phase 3 Study to Assess the Efficacy and Safety of BoNT/A-DP in the Treatment of Glabellar Lines in Comparison With Placebo, Followed by an Open Label Extension Study
Brief Title: Botulinum Toxin Treatment of Glabellar Lines: Efficacy and Safety Study I
Acronym: BLESS I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPH-301-201030; 2015-002164-16 (EudraCT Number)
Record Dates: First submitted 2015-10-22; First posted 2016-02-09 (Estimated); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2022-05

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Botulinum toxin A (Experimental): Botulinum Toxin A (Clostridium botulinum toxin type A) will be administered in double blind fashion in cycle 1. 20 Units will be administered (divided in five 0.1 mL i.m. injections) into the glabellar area.
  Interventions: Drug: Botulinum Toxin A
- Placebo (Placebo Comparator): Placebo will be administered in double blind fashion in cycle 1. divided in five 0.1 mL i.m. injections into the glabellar area.
  Interventions: Drug: Placebo
- Botulinum toxin A Open Label Extension Arm (Experimental): Open Label Extension Arm where all Subjects from Arm 1 and 2 can receive Experimental Treatment in up to 3 treatment cycles.
  20 Units will be administered (divided in five 0.1 mL i.m. injections) into the glabellar area.
  Interventions: Drug: Botulinum Toxin A

INTERVENTIONS:
Drug: Botulinum Toxin A — Injection, 20 Units divided in five 0.1 mL i.m. injections into the glabellar area.
  Other Names: BoNT/A-DP
  Arms: Botulinum toxin A
Drug: Placebo — Injection, 0.9% sodium chloride divided in five 0.1 mL i.m. injections into glabellar area
  Other Names: sodium chloride 0.9%
  Arms: Placebo
Drug: Botulinum Toxin A — Injection, 20 Units divided in five 0.1 mL i.m. injections into the glabellar area in up to 3 treatment cycles
  Other Names: BoNT/A-DP
  Arms: Botulinum toxin A Open Label Extension Arm

SUMMARY:
The aim of this study is to assess the efficacy and safety of BoNT/A-DP in the treatment of glabellar lines in comparison with placebo, including efficacy after repeat treatments and long term safety.

DETAILED DESCRIPTION:
This multicenter Phase 3 study is comprised of two parts. The first part of the study is a randomized, double blind, placebo-controlled, phase which aims to demonstrate efficacy and safety of BoNT/A-DP compared with placebo. The second part is an open label extension phase to evaluate efficacy after repeat treatments and long term safety. Subjects can receive a maximum of four treatment cycles over the duration of the study, a single treatment in the first cycle compared with placebo, and up to three subsequent treatments in the open label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years or older at the time of screening (upper limit 75 years, inclusive).
* Has moderate to severe glabellar frown lines at maximum frown (severity score of 2 or 3 on FWS) as determined by in-clinic assessments by both the investigator and the subject (where: 0= 'none', 1= 'mild', 2= 'moderate', 3= 'severe').
* Subject has a stable medical condition with no uncontrolled systemic disease.
* Female subjects of childbearing potential must test negative for pregnancy and agree to use highly effective birth control during the course of the study. Such methods include for example: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion or vasectomized partner.
* Subjects who wear glasses must be able to adequately self-assess the severity of their glabellar lines (according to the FWS), without glasses obstructing the forehead area.
* The moderate to severe glabellar lines have an important psychological impact on the subject, as indicated by scores >0 on either the Emotional or Functioning subscales of the modified Skindex-16 (GL-QoL).

Exclusion Criteria:

* Previous treatment with any serotype of botulinum toxin for any indication within the 12 months prior to screening, or any planned treatment with botulinum toxin of any serotype for any reason during the trial (other than the investigational treatment).
* Known hypersensitivity to the study medication or its excipients.
* Any medical condition that may place the subject at increased risk due to exposure to botulinum toxin, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, profound atrophy or weakness in the target muscles, or any other condition (at the investigator's discretion) that might interfere with neuromuscular function or contraindicate botulinum toxin therapy.
* Facial laser or light treatment, microdermabrasion, superficial peels or retinoid therapy within the 3 months prior to screening or planned during the study.
* Apart from the procedures specified above, previous treatment with any facial aesthetic procedure in the glabellar area (including chemical peeling, injection with biodegradable fillers,) within 12 months prior to screening or planned during the study.
* Previous insertion of permanent material in the glabellar area or planned during the study.
* Any surgery, or history of surgery, in the glabellar area including surgical removal of the corrugator, procerus or depressor supercili muscles or a combination of these, or scars in the glabellar area, or such surgery planned during the study.
* Active skin disease/infection or irritation at the treatment area.
* Inability to substantially lessen glabellar frown lines even by physically spreading them apart.
* Use of a muscle relaxant within 2 weeks prior to screening or planned during the study.
* Marked facial asymmetry or ptosis of eyelid and/or eyebrow, or current facial palsy or neuromuscular junction disorders as judged by the investigator.
* Pregnant, breastfeeding or planning to become pregnant during the trial.
* Use of prohibited medication including anticholinergic drugs, or drugs which could interfere with neuromuscular function, including aminoglycoside antibiotics and curare-like compounds within 2 weeks prior to screening or planned during the study.
* Planned surgery with general anaesthetic (use of local anaesthetic outside the glabellar area is permitted).
* Participation in another clinical study within one month of screening and throughout the trial.
* Previous participation in another botulinum toxin aesthetic study which involved the treatment of glabellar lines in combination with canthal lines and/or forehead lines in the previous 18 months.
* Chronic drug or alcohol abuse (as per investigator discretion).

Eligibility Criteria for re-treatment: The following criteria MUST be met for re-treatment:

* At time of re-treatment subject does not have relevant changes to their health status from enrollment, which would have prevented subject's entry into the study according to the inclusion and exclusion criteria
* The subject must have been randomized to receive treatment and must have received at least one treatment (BoNT/A-DP or placebo).
* A minimum of 12 weeks must have elapsed since the previous study treatment.
* The subject's glabellar lines at maximum frown must have relapsed to a FWS score of 2 or 3 as determined by the investigator and the subject.
* No relevant infection or inflammation in the planned injection area.
* Negative urine pregnancy test, in women of child-bearing potential.
* The subject must have received fewer than four study treatments.
* The subject must agree and consent to re-treatment.
* Re-treatment will be performed at the latest by week 48.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (9):
  - Total Skin And Beauty Dermatology Center, Pc, Birmingham, Alabama
  - Clinical Testing of Beverly Hills, Encino, California
  - Maas Clinic, San Francisco, California
  - About Skin, Greenwood Village, Colorado
  - DeNova Research, Chicago, Illinois
  - Skin Specialists, Omaha, Nebraska
  - Aesthetic Solutions, Chapel Hill, North Carolina
  - Society Hill Dermatology, Philadelphia, Pennsylvania
  - Tennessee Clinical Research Center, Nashville, Tennessee
- Germany (5):
  - Praxisklinik Fur Dermatologie, Hautzentrum am Starnberger See, Starnberg, Bavaria
  - Rosenpark Research, Darmstadt, Hesse
  - RZANY & HUND, Privatpraxis, Berlin
  - S-thetic Clinic Hamburg, Hamburg
  - Praxis Klinik Dr. Med. Anita Ruetter, Münster
- Poland (4):
  - Carpe Diem, Centre for Aesthetic Medicine, Warsaw
  - Clinical Research Group Sp. z o.o., Warsaw
  - Estederm Dr Marcin Ambroziak, Warsaw
  - High-Med. Przychodnia Specjalistyczna, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox SE, Kaufman-Janette J, Cohen JL, Gold M, Joseph J, Nestor MS, Rzany B, Taylor S, Zhou J, Cecerle M, Pueraro E, Irvine R, Dayan S. LetibotulinumtoxinA Attenuates the Psychological Burden of Glabellar Lines and Is Associated With High Subject Satisfaction in Phase 3 Clinical Trials. Dermatol Surg. 2024 Jun 1;50(6):535-541. doi: 10.1097/DSS.0000000000004152. Epub 2024 Mar 12. PMID 38470985

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 784 enrolled participants, 708 met inclusion criteria and were randomized to treatment.
Groups:
- Botulinum Toxin A Open Label Extension Arm: Open Label Extension Arm where all Subjects from Arm 1 and 2 can receive Experimental Treatment in up to 3 treatment cycles.
  20 Units will be administered (divided in five 0.1 mL i.m. injections) into the glabellar area.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m. injections into the glabellar area in up to 3 treatment cycles
Period: Double Blind Phase
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Started | 531 | 177 | 0
Received Treatment | 529 | 175 | 0
Completed | 502 | 160 | 0
Not Completed | 29 | 17 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Physician Decision | 5 | 0 | 0
Not completed — Lost to Follow-up | 11 | 7 | 0
Not completed — Withdrawal by Subject | 11 | 8 | 0
Not completed — No study drug available at site | 0 | 1 | 0
Period: Open Label Phase
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Started | 0 | 0 | 659 (3 participants who completed the Double-Blind Phase did not enroll into the Open-Label Phase because they were not eligible for retreatment while participating in the study.)
Completed | 0 | 0 | 599
Not Completed | 0 | 0 | 60
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 17
Not completed — Withdrawal by Subject | 0 | 0 | 38

BASELINE CHARACTERISTICS:
Population: The population used consists of all randomized subjects, who received at least one injection with study medication (independent of whether it is BoNT/A-DP or placebo). Participants were analyzed as randomized.
Groups:
- Placebo: Placebo will be administered in double blind fashion in cycle 1. divided in five 0.1 mL i.m. injections into the glabellar area.
  Placebo: Injection, 0.9% sodium chloride divided in five 0.1mL i.m. injections into glabellar area
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin A | Placebo | Total
Number analyzed (Participants) | 529 | 175 | 704
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 463 | 157 | 620
  >=65 years | 66 | 18 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.25 (11.984) | 48.74 (11.378) | 49.13 (11.830)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 463 | 157 | 620
  Male | 66 | 18 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 8 | 33
  Not Hispanic or Latino | 498 | 166 | 664
  Unknown or Not Reported | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 8 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 18 | 51
  White | 482 | 153 | 635
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 269 | 95 | 364
  Germany | 139 | 41 | 180
  Poland | 121 | 39 | 160
Facial Wrinkle Scale at Maximum Frown by Investigator and Subject In-clinic Assessment [Count of Participants; unit: Participants]
  Investigator's In clinic Assessment: No facial wrinkles | 0 | 0 | 0
  Investigator's In clinic Assessment: Mild facial wrinkles | 0 | 0 | 0
  Investigator's In clinic Assessment: Moderate facial wrinkles | 145 | 42 | 187
  Investigator's In clinic Assessment: Severe facial wrinkles | 384 | 133 | 517
  Subject's In-clinic Assessment: No facial wrinkles | 0 | 0 | 0
  Subject's In-clinic Assessment: Mild facial wrinkles | 1 | 0 | 1
  Subject's In-clinic Assessment: Moderate facial wrinkles | 127 | 54 | 181
  Subject's In-clinic Assessment: Severe facial wrinkles | 401 | 121 | 522

OUTCOME MEASURES:

1. Primary Outcome: Facial Wrinkle Scale (FWS) Score of 0 or 1 and an Improvement of ≥ 2 Points in FWS Score (at Maximum Frown) at Week 4 Visit Relative to Baseline, Based on Both the Investigators´ and the Subjects´ In-clinic Assessments.
Description: The primary endpoint is the percentage of subjects among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at week 4 visit (of the first treatment cycle) relative to baseline (responders), based on both the investigators' and the subjects' in-clinic assessments. Thus, the primary endpoint is a composite endpoint comprising investigator and subject assessments of treatment effectiveness. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 4
Population: The population used consists of all randomized subjects, who received at least one injection with study medication. Participants were analyzed as randomized. Participants with missing investigator or subject in-clinic assessments with the Facial Wrinkle Scale (FWS) at baseline or week 4 were assigned as being non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 529 | 175
Participants | 246 | 0
Statistical Analysis 1: Comparison: Botulinum Toxin A vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Responders at Maximum Frown at Week 12
Description: Percentage of subjects among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at week 12 visit (of the first treatment cycle) relative to baseline (responders), based on both the investigators' and the subjects' in-clinic assessments. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 12
Population: The population used consists of all randomized subjects, who received at least one injection with study medication. Participants were analyzed as randomized. Participants with missing investigator or subject in-clinic assessments with the Facial Wrinkle Scale (FWS) at baseline or week 12 were assigned as being non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 529 | 175
Participants | 67 | 0
Statistical Analysis 1: Comparison: Botulinum Toxin A vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — For the testing a hierarchical approach has been applied. The result of this test is considered confirmative if the test of the Primary Outcome Measure shows a confirmatory result at a one-sided significance level of 0.025

3. Secondary Outcome: Percentage of Responders at Week 16
Description: Percentage of subjects among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at week 16 visit (of the first treatment cycle) relative to baseline (responders), based on both the investigators' and the subjects' in-clinic assessments. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 16
Population: The population used consists of all randomized subjects who received at least one injection with study medication and for whom data are available for week 16 or who were re-treated before week 16. They were analyzed as randomized and participants who were re-treated before week 16 were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 501 | 159
Participants | 22 | 0
Statistical Analysis 1: Comparison: Botulinum Toxin A; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel — For the testing a hierarchical approach has been applied. The result of this test is considered confirmative if the test of the Primary and all previous Secondary Outcome Measures show a confirmatory result at a one-sided significance level of 0.025

4. Secondary Outcome: The Percentage of Subjects With a ≥ 1 Point Reduction in Facial Wrinkle Scale (FWS) Score at Rest at Week 4 Based Separately on the Investigators´ and the Subjects´ In-clinic Assessments
Description: The percentage of subjects with a ≥ 1 point reduction in Facial Wrinkle Scale (FWS) score at rest at week 4 in the first treatment cycle, based separately on the investigators' and the subjects' in-clinic assessments (applicable only for subjects who have a FWS score at rest ≥ 1 at baseline). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 4
Population: The population used consists of all randomized subjects who received at least one injection with study medication and who had a Facial Wrinkle Scale (FWS) score at rest >=1 at baseline. Participants were analyzed as randomized. Participants with missing investigator or subject in-clinic assessments with the Facial Wrinkle Scale at week 4 were assigned as being non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 529 | 175
Participants
  Investigator's In-clinic Assessment: number analyzed (Participants) | 474 | 160
  Investigator's In-clinic Assessment | 334 | 27
  Subject's In-clinic Assessment: number analyzed (Participants) | 502 | 167
  Subject's In-clinic Assessment | 412 | 17
Statistical Analysis 1: Comparison: Botulinum Toxin A vs Placebo; Test performed for Investigator's In-clinic Assessment; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Botulinum Toxin A vs Placebo; Test performed for Subject's In-clinic Assessment; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Responders at Week 20 or Later (After the First Treatment).
Description: Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement ≥2 points in FWS score (at maximum frown) at the week 20 visit (or later) relative to baseline, based on both the investigator's and the subject's in-clinic assessment percentage of subjects among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at week 20 visit or later in the first treatment cycle), relative to baseline (responders), based on both the investigators' and the subjects' in-clinic assessments. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 20, 24, 28, 32 of Treatment Cycle 1
Population: The week 20 analysis population includes all randomized subjects who received at least one injection with study medication and have data available or were re-treated before week 20, with re-treated participants counted as non-responders. Post-week 20 analysis includes all randomized subjects with at least one injection with study medication, available data for the respective visit, and no re-treatment before that visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 529 | 175
Participants
  Week 20: number analyzed (Participants) | 503 | 158
  Week 20 | 6 | 0
  Week 24: number analyzed (Participants) | 38 | 1
  Week 24 | 1 | 0
  Week 28: number analyzed (Participants) | 14 | 1
  Week 28 | 0 | 0
  Week 32: number analyzed (Participants) | 12 | 0
  Week 32 | 0 | 0
Statistical Analysis 1: Comparison: Botulinum Toxin A vs Placebo; Test performed for responders rates at week 20; Test type: Superiority; p = 0.084, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Extent of Change in Psychological Impact
Description: Extent of change in psychological impact at week 4 after first treatment, relative to baseline, assessed by modified Skindex-16 (Glabellar Line Quality of Life Scale, [GL-QoL]): Each of 7 items rated on 5-point scale: 0/Never, 1/Rarely, 2/Sometimes, 3/Often, 4/Always bothered, than rescaled to a 0 to 100 standardized score; Emotional Domain is the mean of 4 of the items; Social Functioning Domain is the mean of 3 of the items; Overall score is the mean of all 7 items. All reported scores ranging from 0 (best outcome) to 100 (worst outcome).
  validated FACE-Q Appraisal of Lines Between Eyebrows scale: Each of 7 items rated on 4-point scale: 1/Not at all, 2/a little, 3/moderately, 4/extremely. Reported score is the sum of the 7 items, standardized on a scale from 0 (worst outcome) to 100 (best outcome).
  Age Appraisal visual analog scale [VAS]: Perception of Age compared to actual age, in years ranging from -15 years (best outcome) to +15 years (worst outcome).
Time Frame: Week 4
Population: The population used consists of all randomized subjects, who received at least one injection with study medication and who have data available for week 4. Participants were analyzed as randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 522 | 168
units on a scale
  Modified Skindex-16 (GL-QoL) Emotional domain - Change from Baseline at Week 4 | -32.74 (31.134) | 0.63 (16.997)
  Modified Skindex-16 (GL-QoL) Social Functioning domain - Change from Baseline at Week 4 | -27.44 (30.358) | -1.14 (22.041)
  Modified Skindex-16 (GL-QoL) Overall score - Change from Baseline at Week 4 | -30.47 (28.707) | -0.14 (16.637)
  FACE-Q Appraisal of Lines Between Eyebrows - Change from Baseline at Week 4 | 37.80 (25.917) | -2.05 (14.913)
  Age Appraisal VAS - Change from Baseline at Week 4 | -2.45 (4.531) | -0.27 (3.379)
Statistical Analysis 1: Comparison: Botulinum Toxin A vs Placebo; Test performed for the Modified Skindex-16 (GL-QoL) Emotional domain change from baseline at week 4; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Botulinum Toxin A vs Placebo; This test was performed for the Modified Skindex-16 (GL-QoL) Functioning domain - Change from baseline at Week 4; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Botulinum Toxin A vs Placebo; This test was performed for the Modified Skindex-16 (GL-QoL) Overall score; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Botulinum Toxin A vs Placebo; Test was performed for the FACE-Q Appraisal of Lines Between Eyebrows Scale - Change from Baseline at Week 4; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Botulinum Toxin A vs Placebo; Test was performed for the FACE-Q Age Appraisal VAS score; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Responder Rate at Weeks 1, 2 and 8
Description: The percentage of responders among BoNT/A-DP and placebo groups with a Facial Wrinkle Scale (FWS) score at maximum frown of 0 or 1 and an improvement ≥ 2 points in FWS score (at maximum frown) during the first treatment cycle visit relative to baseline, based on both the investigators' and the subjects' in-clinic assessments (composite endpoint, at weeks 1, 2 and 8). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 1, Week 2, and Week 8
Population: The population used consists of all randomized subjects, who received at least one injection with study medication (independent of whether it is BoNT/A-DP or placebo). Participants were analyzed as randomized. Participants with missing investigator or subject in-clinic assessments with the Facial Wrinkle Scale (FWS) at baseline or the respective visit were assigned as being non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 529 | 175
Participants
  Week 1 | 207 | 0
  Week 2 | 265 | 0
  Week 8 | 152 | 0

8. Secondary Outcome: The Percentage of Subjects With ≥ 2-point Reduction in Facial Wrinkle Scale (FWS) Score (at Maximum Frown)
Description: The percentage of subjects with ≥ 2-point reduction in Facial Wrinkle Scale (FWS) score (at maximum frown) in the BoNT/A-DP and placebo groups during the first treatment cycle visit relative to baseline, based on the independent rater's assessment of photographs (at baseline and visits 2, 4, 12, 16 and 20 weeks after treatment, within the first treatment cycle). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 2, 4, 12, 16 and 20
Population: The population used consists of all randomized subjects, who received at least one injection with study medication and for whom independent rater's assessments of photographs are available for the respective timepoint. Participants were analyzed as randomized. The median of all assessments for the same photograph were taken into account.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 511 | 164
Participants
  Week 2 | 351 | 4
  Week 4: number analyzed (Participants) | 506 | 164
  Week 4 | 323 | 5
  Week 12: number analyzed (Participants) | 301 | 159
  Week 12 | 48 | 2
  Week 16: number analyzed (Participants) | 112 | 1
  Week 16 | 23 | 0
  Week 20: number analyzed (Participants) | 54 | 1
  Week 20 | 11 | 0

9. Secondary Outcome: Time to Onset of Effect in the BoNT/A-DP and Placebo Groups in the First Treatment Cycle
Description: Time to onset of effect in the BoNT/A-DP and placebo groups in the first treatment cycle, as measured at weeks 1, 2 and 4 based separately on subject and investigator assessment. Onset of effect defined as at least a 1 point improvement in Facial Wrinkle Scale (FWS) score from baseline (at maximum frown). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: From treatment at Day 0 to Week 4 in Treatment Cycle 1
Population: The population used consists of all randomized subjects who received at least one injection with study drug. Participants were analyzed as randomized.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 529 | 175
Days | 8.0 [8.0 to 9.0] | NA [NA to NA] — The median and inter-quartile range cannot be calculated due to the low number of subjects showing an effect in this arm.

10. Secondary Outcome: Satisfaction With Treatment, During Each Treatment Cycle, as Assessed by the Validated FACE-Q Satisfaction With Outcome Scale.
Description: The extent of subject perceptions of effect of, and satisfaction with, treatment in the BoNT/A-DP and placebo groups, at week 4 of each treatment cycle, as assessed by the validated FACE-Q Satisfaction with Outcome Scale. The FACE-Q Satisfaction with Outcome scale is a patient-reported outcome measure designed to assess a patient's satisfaction with the results of a facial aesthetic procedure. This scale comprises six items, each with four response options: "definitely agree," "somewhat agree," "somewhat disagree," and "definitely disagree."
Time Frame: Week 4 of Treatment Cycles 1, 2, 3 and 4
Population: The population used consists of all randomized subjects, who received at least one injection with study medication in the respective treatment cycle. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 529 | 175 | 659
Participants
  Cycle 1 Week 4 - pleased: number analyzed (Participants) | 529 | 175 | 0
  Cycle 1 Week 4 - pleased: Definitely disagree | 52 | 143 |
  Cycle 1 Week 4 - pleased: Somewhat disagree | 29 | 9 |
  Cycle 1 Week 4 - pleased: Somewhat agree | 121 | 12 |
  Cycle 1 Week 4 - pleased: Definitely agree | 320 | 4 |
  Cycle 1 Week 4 - pleased: Missing | 7 | 7 |
  Cycle 1 Week 4 - expected: number analyzed (Participants) | 529 | 175 | 0
  Cycle 1 Week 4 - expected: Definitely disagree | 56 | 139 |
  Cycle 1 Week 4 - expected: Somewhat disagree | 51 | 12 |
  Cycle 1 Week 4 - expected: Somewhat agree | 169 | 13 |
  Cycle 1 Week 4 - expected: Definitely agree | 246 | 4 |
  Cycle 1 Week 4 - expected: Missing | 7 | 7 |
  Cycle 1 Week 4 - great: number analyzed (Participants) | 529 | 175 | 0
  Cycle 1 Week 4 - great: Definitely disagree | 59 | 151 |
  Cycle 1 Week 4 - great: Somewhat disagree | 61 | 6 |
  Cycle 1 Week 4 - great: Somewhat agree | 130 | 8 |
  Cycle 1 Week 4 - great: Definitely agree | 272 | 3 |
  Cycle 1 Week 4 - great: Missing | 7 | 7 |
  Cycle 1 Week 4 - look in the mirror: number analyzed (Participants) | 529 | 175 | 0
  Cycle 1 Week 4 - look in the mirror: Definitely disagree | 65 | 146 |
  Cycle 1 Week 4 - look in the mirror: Somewhat disagree | 71 | 10 |
  Cycle 1 Week 4 - look in the mirror: Somewhat agree | 198 | 9 |
  Cycle 1 Week 4 - look in the mirror: Definitely agree | 188 | 3 |
  Cycle 1 Week 4 - look in the mirror: Missing | 7 | 7 |
  Cycle 1 Week 4 - fantastic: number analyzed (Participants) | 529 | 175 | 0
  Cycle 1 Week 4 - fantastic: Definitely disagree | 80 | 152 |
  Cycle 1 Week 4 - fantastic: Somewhat disagree | 72 | 7 |
  Cycle 1 Week 4 - fantastic: Somewhat agree | 164 | 6 |
  Cycle 1 Week 4 - fantastic: Definitely agree | 206 | 3 |
  Cycle 1 Week 4 - fantastic: Missing | 7 | 7 |
  Cycle 1 Week 4 - miraculous: number analyzed (Participants) | 529 | 175 | 0
  Cycle 1 Week 4 - miraculous: Definitely disagree | 107 | 155 |
  Cycle 1 Week 4 - miraculous: Somewhat disagree | 95 | 5 |
  Cycle 1 Week 4 - miraculous: Somewhat agree | 187 | 5 |
  Cycle 1 Week 4 - miraculous: Definitely agree | 133 | 3 |
  Cycle 1 Week 4 - miraculous: Missing | 7 | 7 |
  Cycle 2 Week 4 - pleased: number analyzed (Participants) | 0 | 0 | 659
  Cycle 2 Week 4 - pleased: Definitely disagree |  |  | 40
  Cycle 2 Week 4 - pleased: Somewhat disagree |  |  | 37
  Cycle 2 Week 4 - pleased: Somewhat agree |  |  | 166
  Cycle 2 Week 4 - pleased: Definitely agree |  |  | 398
  Cycle 2 Week 4 - pleased: Missing |  |  | 18
  Cycle 2 Week 4 - expected: number analyzed (Participants) | 0 | 0 | 659
  Cycle 2 Week 4 - expected: Definitely disagree |  |  | 44
  Cycle 2 Week 4 - expected: Somewhat disagree |  |  | 83
  Cycle 2 Week 4 - expected: Somewhat agree |  |  | 159
  Cycle 2 Week 4 - expected: Definitely agree |  |  | 355
  Cycle 2 Week 4 - expected: Missing |  |  | 18
  Cycle 2 Week 4 - great: number analyzed (Participants) | 0 | 0 | 659
  Cycle 2 Week 4 - great: Definitely disagree |  |  | 54
  Cycle 2 Week 4 - great: Somewhat disagree |  |  | 78
  Cycle 2 Week 4 - great: Somewhat agree |  |  | 151
  Cycle 2 Week 4 - great: Definitely agree |  |  | 357
  Cycle 2 Week 4 - great: Missing |  |  | 19
  Cycle 2 Week 4 - look in the mirror: number analyzed (Participants) | 0 | 0 | 659
  Cycle 2 Week 4 - look in the mirror: Definitely disagree |  |  | 55
  Cycle 2 Week 4 - look in the mirror: Somewhat disagree |  |  | 90
  Cycle 2 Week 4 - look in the mirror: Somewhat agree |  |  | 249
  Cycle 2 Week 4 - look in the mirror: Definitely agree |  |  | 247
  Cycle 2 Week 4 - look in the mirror: Missing |  |  | 18
  Cycle 2 Week 4 - fantastic: number analyzed (Participants) | 0 | 0 | 659
  Cycle 2 Week 4 - fantastic: Definitely disagree |  |  | 77
  Cycle 2 Week 4 - fantastic: Somewhat disagree |  |  | 93
  Cycle 2 Week 4 - fantastic: Somewhat agree |  |  | 202
  Cycle 2 Week 4 - fantastic: Definitely agree |  |  | 269
  Cycle 2 Week 4 - fantastic: Missing |  |  | 18
  Cycle 2 Week 4 - miraculous: number analyzed (Participants) | 0 | 0 | 659
  Cycle 2 Week 4 - miraculous: Definitely disagree |  |  | 114
  Cycle 2 Week 4 - miraculous: Somewhat disagree |  |  | 114
  Cycle 2 Week 4 - miraculous: Somewhat agree |  |  | 223
  Cycle 2 Week 4 - miraculous: Definitely agree |  |  | 190
  Cycle 2 Week 4 - miraculous: Missing |  |  | 18
  Cycle 3 Week 4 - pleased: number analyzed (Participants) | 0 | 0 | 616
  Cycle 3 Week 4 - pleased: Definitely disagree |  |  | 36
  Cycle 3 Week 4 - pleased: Somewhat disagree |  |  | 38
  Cycle 3 Week 4 - pleased: Somewhat agree |  |  | 166
  Cycle 3 Week 4 - pleased: Definitely agree |  |  | 347
  Cycle 3 Week 4 - pleased: Missing |  |  | 29
  Cycle 3 Week 4 - expected: number analyzed (Participants) | 0 | 0 | 616
  Cycle 3 Week 4 - expected: Definitely disagree |  |  | 42
  Cycle 3 Week 4 - expected: Somewhat disagree |  |  | 57
  Cycle 3 Week 4 - expected: Somewhat agree |  |  | 180
  Cycle 3 Week 4 - expected: Definitely agree |  |  | 308
  Cycle 3 Week 4 - expected: Missing |  |  | 29
  Cycle 3 Week 4 - great: number analyzed (Participants) | 0 | 0 | 616
  Cycle 3 Week 4 - great: Definitely disagree |  |  | 50
  Cycle 3 Week 4 - great: Somewhat disagree |  |  | 65
  Cycle 3 Week 4 - great: Somewhat agree |  |  | 174
  Cycle 3 Week 4 - great: Definitely agree |  |  | 296
  Cycle 3 Week 4 - great: Missing |  |  | 31
  Cycle 3 Week 4 - look in mirror: number analyzed (Participants) | 0 | 0 | 616
  Cycle 3 Week 4 - look in mirror: Definitely disagree |  |  | 52
  Cycle 3 Week 4 - look in mirror: Somewhat disagree |  |  | 96
  Cycle 3 Week 4 - look in mirror: Somewhat agree |  |  | 221
  Cycle 3 Week 4 - look in mirror: Definitely agree |  |  | 218
  Cycle 3 Week 4 - look in mirror: Missing |  |  | 29
  Cycle 3 Week 4 - fantastic: number analyzed (Participants) | 0 | 0 | 616
  Cycle 3 Week 4 - fantastic: Definitely disagree |  |  | 70
  Cycle 3 Week 4 - fantastic: Somewhat disagree |  |  | 92
  Cycle 3 Week 4 - fantastic: Somewhat agree |  |  | 194
  Cycle 3 Week 4 - fantastic: Definitely agree |  |  | 231
  Cycle 3 Week 4 - fantastic: Missing |  |  | 29
  Cycle 3 Week 4 - miraculous: number analyzed (Participants) | 0 | 0 | 616
  Cycle 3 Week 4 - miraculous: Definitely disagree |  |  | 109
  Cycle 3 Week 4 - miraculous: Somewhat disagree |  |  | 97
  Cycle 3 Week 4 - miraculous: Somewhat agree |  |  | 214
  Cycle 3 Week 4 - miraculous: Definitely agree |  |  | 167
  Cycle 3 Week 4 - miraculous: Missing |  |  | 29
  Cycle 4 Week 4 - pleased: number analyzed (Participants) | 0 | 0 | 464
  Cycle 4 Week 4 - pleased: Definitely disagree |  |  | 30
  Cycle 4 Week 4 - pleased: Somewhat disagree |  |  | 37
  Cycle 4 Week 4 - pleased: Somewhat agree |  |  | 140
  Cycle 4 Week 4 - pleased: Definitely agree |  |  | 254
  Cycle 4 Week 4 - pleased: Missing |  |  | 3
  Cycle 4 Week 4 - expected: number analyzed (Participants) | 0 | 0 | 464
  Cycle 4 Week 4 - expected: Definitely disagree |  |  | 37
  Cycle 4 Week 4 - expected: Somewhat disagree |  |  | 51
  Cycle 4 Week 4 - expected: Somewhat agree |  |  | 159
  Cycle 4 Week 4 - expected: Definitely agree |  |  | 214
  Cycle 4 Week 4 - expected: Missing |  |  | 3
  Cycle 4 Week 4 - great: number analyzed (Participants) | 0 | 0 | 464
  Cycle 4 Week 4 - great: Definitely disagree |  |  | 50
  Cycle 4 Week 4 - great: Somewhat disagree |  |  | 62
  Cycle 4 Week 4 - great: Somewhat agree |  |  | 138
  Cycle 4 Week 4 - great: Definitely agree |  |  | 211
  Cycle 4 Week 4 - great: Missing |  |  | 3
  Cycle 4 Week 4 - look in the mirror: number analyzed (Participants) | 0 | 0 | 464
  Cycle 4 Week 4 - look in the mirror: Definitely disagree |  |  | 41
  Cycle 4 Week 4 - look in the mirror: Somewhat disagree |  |  | 88
  Cycle 4 Week 4 - look in the mirror: Somewhat agree |  |  | 175
  Cycle 4 Week 4 - look in the mirror: Definitely agree |  |  | 157
  Cycle 4 Week 4 - look in the mirror: Missing |  |  | 3
  Cycle 4 Week 4 - fantastic: number analyzed (Participants) | 0 | 0 | 464
  Cycle 4 Week 4 - fantastic: Definitely disagree |  |  | 58
  Cycle 4 Week 4 - fantastic: Somewhat disagree |  |  | 97
  Cycle 4 Week 4 - fantastic: Somewhat agree |  |  | 154
  Cycle 4 Week 4 - fantastic: Definitely agree |  |  | 152
  Cycle 4 Week 4 - fantastic: Missing |  |  | 3
  Cycle 4 Week 4 - miraculous: number analyzed (Participants) | 0 | 0 | 464
  Cycle 4 Week 4 - miraculous: Definitely disagree |  |  | 92
  Cycle 4 Week 4 - miraculous: Somewhat disagree |  |  | 97
  Cycle 4 Week 4 - miraculous: Somewhat agree |  |  | 152
  Cycle 4 Week 4 - miraculous: Definitely agree |  |  | 120
  Cycle 4 Week 4 - miraculous: Missing |  |  | 3

11. Secondary Outcome: The Percentage of Subjects With a ≥ 1 Point Reduction in Facial Wrinkle Scale (FWS) Score at Rest Based on the Independent Rater's Assessment of Photos.
Description: The percentage of subjects with a ≥ 1 point reduction in Facial Wrinkle Scale (FWS) score at rest in the BoNT/A-DP and placebo groups, relative to baseline, during the first treatment cycle, based on the independent rater's assessment of photos. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 2, 4, 12, 16, 20, 24 and 28 of Treatment Cycle 1
Population: The population used consists of all randomized subjects, who received at least one injection with study medication and for whom independent rater's assessments of photographs were performed. Participants were analyzed as randomized. The median of all assessments for the same photograph were taken into account.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo
Number analyzed (Participants) | 529 | 175
Participants
  Week 2: number analyzed (Participants) | 511 | 164
  Week 2 | 184 | 18
  Week 4: number analyzed (Participants) | 506 | 164
  Week 4 | 166 | 19
  Week 12: number analyzed (Participants) | 301 | 159
  Week 12 | 93 | 22
  Week 16: number analyzed (Participants) | 112 | 1
  Week 16 | 30 | 0
  Week 20: number analyzed (Participants) | 54 | 1
  Week 20 | 9 | 1
  Week 24: number analyzed (Participants) | 23 | 1
  Week 24 | 6 | 0
  Week 28: number analyzed (Participants) | 3 | 0
  Week 28 | 1 | 0

12. Secondary Outcome: Facial Wrinkle Scale (FWS) Score of 0 or 1 and an Improvement of ≥ 2 Points in FWS Score (at Maximum Frown) at 4 Weeks After Re-treatment Relative to the Rating at the Preceding End-of-Cycle Visit.
Description: The percentage of subjects with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at 4 weeks after re-treatment relative to the rating at the preceding end-of-cycle visit, based on both the investigator's and the subject's in-clinic assessments (composite endpoint). FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles.
Time Frame: Week 4 of Treatment Cycles 2, 3 and 4
Population: The population used consists of all randomized subjects who received at least one injection with study medication and for whom data are available for the respective timepoint. Participants were analyzed as randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 659
Participants
  Week 4 after 1st Re-treatment: number analyzed (Participants) | 639
  Week 4 after 1st Re-treatment | 245
  Week 4 after 2nd Re-treatment: number analyzed (Participants) | 587
  Week 4 after 2nd Re-treatment | 187
  Week 4 after 3rd Re-treatment: number analyzed (Participants) | 462
  Week 4 after 3rd Re-treatment | 104

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious AEs (SAEs) and Adverse Events of Special Interest (AESIs) Events of Special Interest (AESIs)
Description: Frequency, severity and causal relationship of adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) during the entire study period.
Time Frame: Through study completion (60 weeks)
Population: The population used consists of all randomized subjects, who received at least one injection with study medication. Participants were analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 529 | 175 | 659
Participants
  Subjects with any Treatment Emergent Adverse Event (TEAE) | 129 | 39 | 268
  Subjects with any Study Medication Related TEAE | 19 | 4 | 31
  Subjects with any Injection Procedure Related TEAE | 22 | 8 | 29
  Subjects with any Severe TEAE | 12 | 3 | 17
  Subjects with any Serious TEAE | 9 | 0 | 15
  Subjects with any Adverse Events of Special Interest (AESI) | 1 | 1 | 3

14. Secondary Outcome: Number of Participants With Neutralizing Anti-Drug Antibodies
Description: Number of Participants with Neutralizing Anti-Drug Antibodies Antibody formation, evaluation pre-dose before each treatment, at 4 weeks after each treatment and at the final study visit
Time Frame: Through study completion (60 weeks)
Population: The population used consists of all subjects who received at least one injection with study medication. Participants were analyzed as treated. Confirmation assays have only been performed for subjects with a reactive Screening Assay result.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
Number analyzed (Participants) | 529 | 175 | 659
Participants
  Baseline - Anti-Drug Antibodies (ADA) Screening Assay - Reactive: number analyzed (Participants) | 529 | 175 | 0
  Baseline - Anti-Drug Antibodies (ADA) Screening Assay - Reactive | 37 | 11 |
  Baseline - ADA Confirmation Assay - Confirmed: number analyzed (Participants) | 37 | 11 | 0
  Baseline - ADA Confirmation Assay - Confirmed | 3 | 0 |
  End of Study - ADA Screening Assay - Reactive: number analyzed (Participants) | 0 | 0 | 659
  End of Study - ADA Screening Assay - Reactive |  |  | 64
  End of Study - ADA Confirmation Assay - Confirmed: number analyzed (Participants) | 0 | 0 | 64
  End of Study - ADA Confirmation Assay - Confirmed |  |  | 2

15. Secondary Outcome: Change From Baseline of Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase
Description: Safety assessments by evaluating change from baseline of Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: The population used consists of all subjects who received at least one injection with study medication and have data available for the respective visit. Participants were analyzed as treated.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Botulinum Toxin A: Botulinum Toxin A will be administered in double blind fashion in Treatment Cycle 1. 20 Units will be administered (divided in five 0.1 mL i.m injections) into glabellar area.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area
- Placebo: Placebo will be administered in double blind fashion in Treatment Cycle 1 divided in five 0.1 mL injections into the glabellar area.
  Placebo: injection, 0.9% sodium chloride divided in five 0.1 mL i.m injections into the glabellar area
- Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2: Open Label Extension Arm where all Subjects from Arm 1 and 2 can receive Experimental Treatment in up to three additional treatment cycles. This arm is designated for Study Treatment Cycle 2.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area in Treatment Cycle 2
- Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3: Open Label Extension Arm where all Subjects from Arm 1 and 2 can receive Experimental Treatment in up to three additional treatment cycles. This arm is designated for Study Treatment Cycle 3.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area in Treatment Cycle
- Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4: Open Label Extension Arm where all Subjects from Arm 1 and 2 can receive Experimental Treatment in up to three additional treatment cycles. This arm is designated for Study Treatment Cycle 4.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area in Treatment Cycle 4
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 516 | 165 | 628 | 577 | 441
U/L
  Week 4 of each treatment cycle - Alanine Aminotransferase (U/L): number analyzed (Participants) | 515 | 163 | 627 | 576 | 439
  Week 4 of each treatment cycle - Alanine Aminotransferase (U/L) | 0.10 (8.091) | -0.34 (14.568) | 0.23 (7.710) | 0.38 (9.788) | 1.09 (12.995)
  Week 4 of each treatment cycle - Alkaline Phosphatase (U/L) | 0.26 (7.667) | -0.19 (10.546) | 1.07 (11.027) | 1.54 (9.698) | 0.42 (9.937)
  Week 4 of each treatment cycle - Aspartate Aminotransferase (U/L): number analyzed (Participants) | 495 | 159 | 624 | 577 | 440
  Week 4 of each treatment cycle - Aspartate Aminotransferase (U/L) | 0.82 (8.501) | 0.56 (8.270) | -0.29 (8.323) | 0.06 (13.801) | -0.04 (9.123)
  Week 4 of each treatment cycle - Gamma Glutamyl Transferase (U/L) | 0.18 (8.991) | 0.01 (10.361) | 0.16 (7.442) | 0.94 (11.723) | 1.62 (11.030)

16. Secondary Outcome: Change From Baseline of Bilirubin and Creatinine
Description: Safety assessments by evaluating change from baseline of Bilirubin and Creatinine as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 516 | 165 | 628 | 577 | 441
μmol/L
  Week 4 of each treatment cycle - Bilirubin (μmol/L): number analyzed (Participants) | 515 | 163 | 627 | 576 | 439
  Week 4 of each treatment cycle - Bilirubin (μmol/L) | 0.28 (3.576) | 0.31 (3.644) | -0.13 (3.221) | -0.30 (3.292) | 0.04 (3.488)
  Week 4 of each treatment cycle - Creatinine (μmol/L) | 0.81 (7.548) | -0.37 (7.465) | 0.09 (8.718) | -0.37 (8.368) | -1.26 (9.450)

17. Secondary Outcome: Change From Baseline of Blood Urea Nitrogen, Cholesterol, Glucose, Potassium, Sodium
Description: Safety assessments by evaluating change from baseline of Blood Urea Nitrogen, Cholesterol, Glucose, Potassium, Sodium as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 516 | 165 | 628 | 577 | 441
mmol/L
  Week 4 of each treatment cycle - Blood Urea Nitrogen (mmol/L) | 0.05 (1.248) | -0.20 (1.151) | -0.04 (1.213) | -0.03 (1.122) | -0.07 (1.257)
  Week 4 of each treatment cycle - Cholesterol (mmol/L) | -0.06 (0.621) | -0.04 (0.614) | 0.03 (0.593) | 0.02 (0.651) | 0.01 (0.677)
  Week 4 of each treatment cycle - Glucose (mmol/L) | 0.05 (1.140) | -0.13 (1.056) | 0.06 (1.168) | 0.06 (1.200) | 0.13 (1.073)
  Week 4 of each treatment cycle - Potassium (mmol/L): number analyzed (Participants) | 503 | 163 | 628 | 577 | 441
  Week 4 of each treatment cycle - Potassium (mmol/L) | 0.03 (0.431) | 0.01 (0.369) | 0.00 (0.387) | 0.01 (0.395) | 0.01 (0.0427)
  Week 4 of each treatment cycle - Sodium (mmol/L) | -0.18 (2.117) | -0.30 (2.013) | 0.14 (2.290) | 0.26 (2.432) | 0.29 (3.150)

18. Secondary Outcome: Change From Baseline of Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Safety assessments by evaluating change from baseline of Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: (x10^9 cells/L)
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 514 | 162 | 622 | 565 | 425
(x10^9 cells/L)
  Week 4 of each treatment cycle - Basophils (x10^9 cells/L): number analyzed (Participants) | 512 | 162 | 620 | 565 | 425
  Week 4 of each treatment cycle - Basophils (x10^9 cells/L) | 0.00 (0.034) | 0.00 (0.036) | 0.00 (0.044) | 0.00 (0.043) | 0.00 (0.043)
  Week 4 of each treatment cycle - Eosinophils (x10^9 cells/L): number analyzed (Participants) | 512 | 162 | 620 | 565 | 425
  Week 4 of each treatment cycle - Eosinophils (x10^9 cells/L) | 0.00 (0.077) | 0.00 (0.058) | 0.02 (0.174) | 0.02 (0.096) | 0.01 (0.094)
  Week 4 of each treatment cycle - Leukocytes (x10^9 cells/L) | -0.22 (1.370) | -0.02 (1.334) | -0.04 (1.560) | -0.01 (1.586) | 0.00 (1.652)
  Week 4 of each treatment cycle - Lymphocytes (x10^9 cells/L): number analyzed (Participants) | 512 | 162 | 620 | 565 | 425
  Week 4 of each treatment cycle - Lymphocytes (x10^9 cells/L) | -0.06 (0.429) | -0.03 (0.481) | 0.03 (0.518) | 0.04 (0.498) | 0.01 (0.451)
  Week 4 of each treatment cycle - Monocytes (x10^9 cells/L): number analyzed (Participants) | 512 | 162 | 620 | 565 | 425
  Week 4 of each treatment cycle - Monocytes (x10^9 cells/L) | 0.00 (0.122) | 0.00 (0.135) | -0.01 (0.125) | -0.02 (0.156) | -0.01 (0.150)
  Week 4 of each treatment cycle - Neutrophils (x10^9 cells/L): number analyzed (Participants) | 512 | 162 | 620 | 565 | 425
  Week 4 of each treatment cycle - Neutrophils (x10^9 cells/L) | -0.16 (1.209) | 0.02 (1.091) | -0.09 (1.310) | -0.06 (1.381) | -0.01 (1.456)
  Week 4 of each treatment cycle - Platelets (x10^9 cells/L): number analyzed (Participants) | 509 | 159 | 620 | 562 | 423
  Week 4 of each treatment cycle - Platelets (x10^9 cells/L) | -4.83 (34.695) | -1.39 (37.755) | 3.91 (32.882) | 6.75 (42.930) | 6.40 (40.506)

19. Secondary Outcome: Change From Baseline of Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes, Neutrophils/Leukocytes
Description: Safety assessments by evaluating change from baseline of Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes, Neutrophils/Leukocyte as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: % of leukocytes
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 512 | 162 | 620 | 565 | 425
% of leukocytes
  Week 4 of each treatment cycle - Basophils/Leukocytes (%) | 0.04 (0.513) | 0.02 (0.532) | -0.02 (0.641) | 0.00 (0.589) | 0.08 (0.660)
  Week 4 of each treatment cycle - Eosinophils/Leukocytes (%) | 0.05 (1.140) | -0.01 (0.920) | 0.27 (1.697) | 0.34 (1.587) | 0.21 (1.594)
  Week 4 of each treatment cycle - Lymphocytes/Leukocytes (%) | 0.12 (6.262) | -0.32 (5.969) | 0.78 (6.390) | 1.06 (7.082) | 0.32 (7.219)
  Week 4 of each treatment cycle - Monocytes/Leukocytes (%) | 0.20 (1.784) | -0.17 (1.890) | -0.07 (1.803) | -0.19 (2.098) | -0.25 (1.958)
  Week 4 of each treatment cycle - Neutrophils/Leukocytes (%) | -0.39 (7.292) | 0.47 (6.890) | -0.96 (7.613) | -1.20 (8.249) | -0.37 (8.321)

20. Secondary Outcome: Change From Baseline of Erythrocytes
Description: Safety assessments by evaluating change from baseline of Erythrocytes as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: (x10^12 cells/L)
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 514 | 162 | 622 | 565 | 425
(x10^12 cells/L) | -0.01 (2.229) | -0.01 (0.210) | 0.02 (0.216) | 0.01 (0.229) | -0.01 (0.211)

21. Secondary Outcome: Change From Baseline of Erythrocytes MCHC, Hemoglobin
Description: Safety assessments by evaluating change from baseline of Erythrocytes MCHC, Hemoglobin as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 514 | 162 | 622 | 565 | 425
g/dL
  Week 4 of each treatment cycle - Erythrocytes MCHC Concentration (g/dL) | -0.17 (1.103) | -0.14 (1.064) | 0.12 (1.139) | -0.03 (1.233) | -0.55 (1.309)
  Week 4 of each treatment cycle - Hemoglobin (g/dL) | -0.01 (0.668) | -0.02 (0.577) | 0.05 (0.627) | -0.03 (0.628) | -0.12 (0.635)

22. Secondary Outcome: Change From Baseline of Erythrocyte MCV
Description: Safety assessments by evaluating change from baseline of Erythrocyte MCV as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 514 | 162 | 622 | 565 | 425
fL | 0.57 (2.968) | 0.49 (2.978) | -0.42 (2.722) | -0.32 (3.472) | 1.08 (4.066)

23. Secondary Outcome: Change From Baseline of Systolic and Diastolic Blood Pressure
Description: Safety assessments by evaluating change from baseline of Systolic and Diastolic Blood Pressure as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 520 | 168 | 640 | 582 | 445
mmHg
  Week 4 of each treatment cycle - Systolic Blood Pressure (mmHg) | -0.70 (12.709) | -1.42 (12.665) | 0.00 (13.136) | 0.00 (12.497) | -0.33 (13.586)
  Week 4 of each treatment cycle - Diastolic Blood Pressure (mmHg) | -0.46 (9.086) | 0.49 (9.574) | 0.60 (8.960) | 0.83 (9.437) | 0.36 (9.525)

24. Secondary Outcome: Change From Baseline of Pulse Rate
Description: Safety assessments by evaluating change from baseline of Pulse Rate as per the study schedule
Time Frame: Week 4 after treatment in treatment cycle 1, 2, 3 and 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 2 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 3 | Botulinum Toxin A Open Label Extension Arm - Treatment Cycle 4
Number analyzed (Participants) | 520 | 168 | 640 | 582 | 445
bpm | -1.24 (9.592) | -0.35 (9.076) | 1.35 (9.002) | 1.54 (9.752) | 1.81 (9.970)

25. Secondary Outcome: Number of Participants With Normal and Abnormal Electrocardiogram
Description: Safety assessments by evaluating Electrocardiogram as per the study schedule
Time Frame: Last visit of Treatment Cycle 1 (End of Cycle procedures) conducted upon confirmation of eligibility for retreatment, which was assessed starting 12 weeks post-treatment with 4-weekly evaluations up to a maximum of 48 weeks post treatment.
Population: The population used consists of all subjects who received at least one injection with study medication and who have data available post baseline and the respective category of baseline electrocardiogram interpretation. Participants were analyzed as treated.
Measure: Count of Participants; unit: Participants
Groups:
- Botulinum Toxin A - Normal Baseline Electrocardiogram Interpretation: Botulinum Toxin A (Clostridium botulinum toxin type A) will be administered in double blind fashion in cycle 1. 20 Units will be administered (divided in five 0.1 mL i.m. injections) into the glabellar area.
  Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m. injections into the glabellar area.
  Subjects had an electrocardiogram interpretation of normal at baseline.
- Botulinum Toxin A - Abnormal Baseline Electrocardiogram Interpretation: Botulinum Toxin A will be administered in double blind fashion in Treatment Cycle 1. 20 Units will be administered (divided in five 0.1 mL i.m injections) into glabellar area. Botulinum Toxin A: Injection, 20 Units divided in five 0.1 mL i.m injections into the glabellar area Subjects had an electrocardiogram interpretation of abnormal at baseline.
- Placebo - Normal Baseline Electrocardiogram Interpretation: Placebo will be administered in double blind fashion in cycle 1. divided in five 0.1 mL i.m. injections into the glabellar area.
  Placebo: Injection, 0.9% sodium chloride divided in five 0.1mL i.m. injections into glabellar area
  Subjects had an electrocardiogram interpretation of normal at baseline.
- Placebo - Abnormal Baseline Electrocardiogram Interpretation: Placebo will be administered in double blind fashion in Treatment Cycle 1 divided in five 0.1 mL injections into the glabellar area.
  Placebo: injection, 0.9% sodium chloride divided in five 0.1 mL i.m injections into the glabellar area
  Subjects had an electrocardiogram interpretation of abnormal at baseline.
Arm/Group | Botulinum Toxin A - Normal Baseline Electrocardiogram Interpretation | Botulinum Toxin A - Abnormal Baseline Electrocardiogram Interpretation | Placebo - Normal Baseline Electrocardiogram Interpretation | Placebo - Abnormal Baseline Electrocardiogram Interpretation
Number analyzed (Participants) | 340 | 174 | 106 | 59
Participants
  Last observation in Cycle 1 - Normal | 280 | 71 | 90 | 25
  Last observation in Cycle 1 - Abnormal | 60 | 103 | 16 | 34

ADVERSE EVENTS:
Time Frame: Up to 60 weeks post first treatment
Arm/Group | Botulinum Toxin A | Placebo | Botulinum Toxin A Open Label Extension Arm
All-Cause Mortality (participants affected / at risk) | 0/529 | 0/175 | 0/659
Serious Adverse Events (participants affected / at risk) | 9/529 | 0/175 | 15/659
Other Adverse Events (participants affected / at risk) | 48/529 | 11/175 | 133/659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin A (N=529) | Placebo (N=175) | Botulinum Toxin A Open Label Extension Arm (N=659)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cervicitis cystic (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin A (N=529) | Placebo (N=175) | Botulinum Toxin A Open Label Extension Arm (N=659)
Influenza (Infections and infestations) | 4 (4) | 3 (3) | 14 (14)
Sinusitis (Infections and infestations) | 6 (6) | 1 (1) | 15 (17)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 17 (17)
Viral upper respiratory tract infection (Infections and infestations) | 23 (23) | 6 (6) | 77 (98)
Headache (Nervous system disorders) | 16 (16) | 1 (1) | 21 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02677298/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT02677298/SAP_001.pdf